CLINICAL TRIAL: NCT05321017
Title: Can Increasing Motor Evoked Potential Size Improve Upper Extremity Motor Function in Individuals With Incomplete Spinal Cord Injury?
Brief Title: Wrist Extensor MEP Up-conditioning for Individuals With Incomplete Spinal Cord Injury
Acronym: uMEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Blair Dellenbach, Occupational Therapist, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00113108
Record Dates: First submitted 2022-03-04; First posted 2022-04-11 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injuries; Quadriplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MEP Wrist Extensor Up-Conditioning (Experimental)
  Interventions: Behavioral: MEP Operant Up-conditioning of the Wrist Extensor

INTERVENTIONS:
Behavioral: MEP Operant Up-conditioning of the Wrist Extensor — This is a training intervention in which the brain-spinal cord-muscle pathways are strengthened in individuals with incomplete spinal cord injury. Transcranial magnetic stimulation (TMS), a type of brain stimulation, will be used to elicit a muscle response from the wrist extensor (extensor carpi radialis), the muscle the bends the wrist back.

SUMMARY:
The purpose of this study is to examine the relationship between common clinical assessments and measurements of the function of brain-spinal cord-muscle connections, and to examine the effects of training a brain-spinal cord-muscle response in individuals with incomplete spinal cord injury. A transcranial magnetic stimulator (TMS) is used for examining brain-to-muscle pathways. This stimulator produces a magnetic field for a very short period of time and indirectly stimulates brain cells with little or no discomfort. The target muscle is the wrist extensor (extensor carpi radialis) muscle that bends the wrist back. It is hypothesized that training the wrist extensor muscle response to transcranial magnetic stimulation will increase the strength of the brain-to-muscle pathway, which will improve the ability to move the arm.

It is hoped that the results of this training study will help in developing therapy strategies for individuals, promoting better understanding of clinical assessments, and understanding treatments that aim to improve function recovery in people with spinal cord injury (SCI).

This study requires 30 visits, and each visit will last approximately 1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

1. a history of injury to spinal cord at or above C6
2. neurologically stable (>6 mo post SCI)
3. medical clearance to participate
4. weak wrist extension at least unilaterally
5. expectation that current medication will be maintained without change for at least 3 months. Stable use of anti-spasticity medication (e.g., baclofen, diazepam, tizanidine) is accepted. In participants with bilateral wrist extension weakness, the more severely impaired arm is studied.

Exclusion Criteria:

1. motoneuron injury
2. medically unstable condition
3. cognitive impairment
4. a history of epileptic seizures
5. metal implants in the cranium
6. implanted biomedical device in or above the chest (e.g., a cardiac pacemaker, cochlear implant)
7. no measurable MEP elicited in the ECR
8. unable to produce any voluntary ECR EMG activity
9. extensive use of functional electrical stimulation to the arm on a daily basis
10. pregnancy (due to changes in posture and potential medical instability).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the excitability/strength of the brain-spinal cord-muscle pathway at the brain level as measured by the Motor Evoked Potential | Baseline and final training session (approximately 2.5 months)
  An increased average MEP size (mV) would indicate increased excitability/strength of the brain-spinal cord-muscle pathway
Change in ability to move the arm as measured by the Action Research Arm Test (ARAT). Maximum score of 57 points | change from baseline to immediately after completing the training protocol
  An increase in ARAT score indicates an improvement in the ability to move the arm
Change in ability to move the arm as measured by the Fugl-Meyer Assessment (FMA) | change from baseline to immediately after completing the training protocol
  An increase in the FMA score indicates better movement of the arm. Maximum score of 66 points
Change in gross manual dexterity as measured by the Box and Block Test (BBT) | change from baseline to immediately after completing the training protocol
  An increased number of blocks moved in 60s indicates increased gross manual dexterity
Change in fine motor ability and finger dexterity as measured by the Nine Hole Peg Test | change from baseline to immediately after completing the training protocol
  Decreased amount of time (s) to place and remove pegs in a peg board indicates improved fine motor ability and finger dexterity
Change in strength as measured by Manual Muscle Testing (MMT) | change from baseline to immediately after completing the training protocol
  Increased score on MMT indicates increased strength in the muscle being tested. The examiner grades the patient's strength on a 0 to 5 scale. 0: No muscle activation; 1: Trace muscle activation, such as a twitch, without achieving full range of motion; 2: Muscle activation with gravity eliminated, achieving full range of motion; 3: Muscle activation against gravity, full range of motion; 4: Muscle activation against some resistance, full range of motion; 5: Muscle activation against examiner's full resistance, full range of motion.
Change in sensation on the back and palm of the hand as measured by the Semmes Weinstein Monofilament Test | change from baseline to immediately after completing the training protocol
  Ability to detect increasingly thinner monofilaments indicates increased sensation
Change in spasticity as measured by the Modified Ashworth Scale (mAS) | change from baseline to immediately after completing the training protocol
  The mAS score ranges from 0: normal muscle tone to 4: rigid in flexion or extension. A decrease in mAS indicates decreased spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Blair Dellenbach, MSOT, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No